CLINICAL TRIAL: NCT02656394
Title: Amelioration of Adverse Ocular Side Effects of Glaucoma Medications in Glaucoma Patients Using Topical GL101 - Proof of Concept, Safety, and Efficacy Study
Brief Title: Amelioration of Adverse Ocular Side Effects of Glaucoma Medications in Glaucoma Patients Using Topical GL101
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Glia, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GL-1
Record Dates: First submitted 2016-01-08; First posted 2016-01-15 (Estimated); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Ocular Surface Disease
Keywords: ocular surface disease; glaucoma medications

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GL101 (Active Comparator): GL101 topical gel
  Interventions: Drug: GL101
- Placebo (Placebo Comparator): Placebo topical gel
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GL101 — Topical Gel
  Other Names: Pro-Ocular
  Arms: GL101
Drug: Placebo — Placebo topical gel
  Arms: Placebo

SUMMARY:
To evaluate the safety and efficacy of 0.5% GL101 topical gel administered twice daily for 28 days in ameliorating adverse ocular side effects in patients under ongoing treatment with glaucoma medications.

DETAILED DESCRIPTION:
The study is to assess the safety and efficacy of a new treatment for ocular surface disease associated with the use of glaucoma medications.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of any race, at least 18 years of age at Visit 1 Screening.
2. Has provided verbal and written informed consent.
3. Be able and willing to follow instructions, including participation in all study assessments and visits.
4. Currently being treated for glaucoma using at least two medications, and be willing to continue on the same regime.
5. Suffers from at least two of the symptoms in the GLIA™ Glaucoma Medication Ocular Side Effect Symptoms Questionnaire at a severity of 2 (moderate) or more.
6. If a woman of childbearing potential, have a negative urine pregnancy test at Visit 1 and be using an adequate method of birth control throughout the study period.

Exclusion Criteria:

1. Comorbidity with other severe or chronic eye conditions that in the judgment of the investigator will interfere with study assessments, such as corneal opacities and scars, dystrophies, epithelial scarring, infections, blood clots, etc.
2. Best corrected visual acuity (BCVA) at baseline <20/200.
3. Has a condition or history that, in the opinion of the investigator, may interfere significantly with the subject's participation in the study.
4. A woman who is pregnant, nursing an infant, or planning a pregnancy.
5. Has a known adverse reaction and/or sensitivity to the study drug or its components.
6. Routine use (more than twice a week) of a chlorinated swimming pool.
7. Unwilling or unable to cease using the following medications during the study period: Topical ocular cyclosporine (e.g. Restasis®), anti-histamines, antipsychotics, or eye gels.
8. Currently enrolled in an investigational drug or device study or have used an investigational drug or device within 30 days prior to Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-01-22 (Actual); Primary Completion 2017-12-04 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Glaucoma medication ocular side effect symptoms | Day 1 to 4 weeks
  Glaucoma medication ocular side effect symptoms:
  * Ocular discomfort
  * Burning
  * Stinging
  * Conjunctival redness
  * Itching
  * Dryness
  * Foreign object sensation
  * Grittiness
  * Pain
  * Eyelid swelling
  * Eyelid redness
  * Photophobia
  * Excessive tearing
  * Crusty lids
  * Blurred vision

SECONDARY OUTCOMES:
Glaucoma medication ocular side effect signs | Day 1 to 4 weeks
  Glaucoma medication ocular side effect signs:
  * Tearscope tear film examination
  * Tear meniscus height (TMH)
  * Tear film break up time (NIKBUT)
  * Bulbar redness (BR)
  * Meibography
  * Conjunctival redness (hyperemia)
  * Blepharitis
  * Lid margin vessel inflammation
  * Punctate keratitis
  * Corneal staining
  * Conjunctival staining
Other signs | Day 1 to 4 weeks
  Other signs:
  * Visual acuity
  * Intraocular pressure
  * Artificial tear use
  * Glaucoma medication compliance

OTHER OUTCOMES:
Adverse events | Day 1 to 4 weeks
  Adverse events:
  * Visual acuity
  * Slit lamp biomicroscopy
  * Undilated fundoscopy examination
  * Intraocular pressure

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ritch, MD, Principal Investigator — New York Eye & Ear Infirmary of Mount Sinai
Locations (1):
- New York Eye & Ear Infirmary of Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided